CLINICAL TRIAL: NCT00046644
Title: Leukotriene Polymorphisms and Montelukast Response - Ancillary to LoDo Trial
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1189; R01HL071394 (NIH)
Record Dates: First submitted 2002-09-30; First posted 2002-10-01 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To elucidate the mechanisms underlying inter-patient variation in response to montelukast, a drug for asthma.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a common disease caused by a complex interaction between genetic and environmental factors. Asthma afflicts 17 million Americans. In 1999, more than 5000 persons died from asthma. Given the significant mortality and morbidity associated with asthma, it is important to continue to develop new strategies for intervention. Leukotriene antagonists are thought to be the most innovative approach to asthma therapy in 20 years. Despite their demonstrated efficacy, safety and popularity, the leukotriene antagonists are associated with a significant degree of inter-patient variability in response, which can limit their safety, efficacy and cost-effectiveness. Several polymorphisms in leukotriene pathway genes can contribute to variability in response. The project will determine if polymorphisms in genes encoding 5-lipoxygenase, leukotriene A4hydrolase, LTC4 synthase, multi-drug resistance protein 1 (MRP1) and LT1 receptor proteins are determinants of response to montelukast treatment.

The study is in response to an Request for Applications entitled Ancillary Studies in Heart, Lung, and Blood Disease Trials which was released by the NHLBI in June 2000 to conduct mechanistic studies in clinical trials related to heart, lung and blood diseases. Specifically, this initiative focuses on the utilization of patients and patient materials from such trials to study the mechanisms underlying the interventions, the mechanisms of disease pathogenesis, surrogate markers or biomarkers of disease activity and therapeutic effect and the mechanisms of human cardiopulmonary and hematologic function. Studies aimed at accelerating the development of new technologies within the context of the mechanistic investigations are also encouraged.

DESIGN NARRATIVE:

DNA will be collected from patients participating in a parent clinical trial entitled: Effectiveness of Low Dose Theophylline as Add-On Therapy in the Treatment of Asthma (LoDo Trial). 627 patients from 19 Asthma Clinical Research Centers will be randomly assigned to receive placebo, or low dose theophylline (300 mg/day) or montelukast, 10 mg daily, for 6 months. Stepwise Linear and Poisson regressions will be performed on outcomes including treatment and genetic covariates, and interaction terms between treatment arm and genetic makeup. Polymorphisms that are highly associated with response can lead to the development of genetic tests that will identify patients most likely to benefit from montelukast treatment. This information may lead to individualization of asthma medications based on the genetic make-up of the patient.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lima — Nemours Children's Clinic

REFERENCES:
- [Derived] Duan QL, Gaume BR, Hawkins GA, Himes BE, Bleecker ER, Klanderman B, Irvin CG, Peters SP, Meyers DA, Hanrahan JP, Lima JJ, Litonjua AA, Tantisira KG, Liggett SB. Regulatory haplotypes in ARG1 are associated with altered bronchodilator response. Am J Respir Crit Care Med. 2011 Feb 15;183(4):449-54. doi: 10.1164/rccm.201005-0758OC. Epub 2010 Sep 17. PMID 20851928